CLINICAL TRIAL: NCT01468636
Title: A Randomized Controlled Trial to Examine the Effectiveness of 400 mg of Oral Zinc Gluconate as Adjunctive Therapy for Ano-genital Warts
Brief Title: A RTC to Examine the Effectiveness of 400 mg of Oral Zinc Gluconate as Adjunctive Therapy for Ano-genital Warts
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: There was no clear benefit but numerous side effects.
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Centre for Disease Control (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H11-01758; H11-01758 (Other: UBC IRB number)
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Genital Warts; HPV
Keywords: Warts; HPV; Zinc
MeSH Terms: conditions — Condylomata Acuminata; Warts | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Zinc (Active Comparator)
  Interventions: Drug: Oral Zinc
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Zinc — 200 mg BID of oral zinc gluconate x 8 weeks
  Arms: Oral Zinc
Drug: Placebo — 200mg BID x 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of 400 mg of oral zinc gluconate on genital warts. Our hypothesis is that there will be a 10% difference in complete clearance of genital warts in the group randomized to oral plus standard of care compared to those randomized to placebo plus standard of care.

DETAILED DESCRIPTION:
Clients presenting to the BCCDC STI clinic with genital warts will be randomized to either 400 mg zinc gluconate or placebo (200mg BID) for 8 weeks in addition to the standard of care. Clinical assessment of warts and additional standard treatment will occur every 7-10 days for a maximum of 8 weeks. A telephone call will occur at week 20 to determine if any of the warts have cleared or re-appeared. The appearance of new warts will also be noted. The proportion of subjects who have complete clearance of genital warts at 8 weeks will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 19 and over
2. Clinical diagnosis of genital warts requiring treatment based on clinician evaluation
3. Fluency in English
4. Available within four days of the intended 8 week follow-up visit

Exclusion Criteria:

1. Individuals under the age of 19
2. Pregnant women
3. Known contraindication to zinc Signs of copper/iron deficiency which include anemia and neutropenia which are characterized by tiredness, fatigue and light headedness.
4. Diseases that alter zinc metabolism or absorption eg. type II diabetes mellitus, Crohn's disease, chronic leg ulcers
5. Clients who are currently taking zinc for therapeutic purposes or have taken zinc in the last two months for therapeutic purposes
6. Clients who have received standard of care treatment for their warts in the past month

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
complete clearance of genital warts | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lester, Principal Investigator — University of British Columbia
Locations (1):
- BC Centre for Disease Control, Vancouver, British Columbia, Canada